CLINICAL TRIAL: NCT02734290
Title: A Pilot and Phase II Study to Assess the Safety, Tolerability and Efficacy of Pembrolizumab Plus Chemotherapy in Metastatic Triple Negative Breast Cancer Patients
Brief Title: Standard of Care Chemotherapy Plus Pembrolizumab for Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-001
Record Dates: First submitted 2016-03-28; First posted 2016-04-12 (Estimated); Results first posted 2024-02-22 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Triple Negative Breast Cancer
Keywords: metastatic; Human epidermal growth factor receptor 2 (HER2) negative breast cancer; Estrogen Receptor (ER) negative breast cancer; Progesterone Receptor (PR) negative breast cancer; Immunotherapy; Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm Metastasis; Breast Neoplasms | interventions — pembrolizumab; Paclitaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): pembrolizumab + weekly paclitaxel
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel
- Arm B (Experimental): pembrolizumab + capecitabine
  Interventions: Drug: Pembrolizumab; Drug: Capecitabine

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg every 3 weeks by IV infusion on Day 1 of each 3 week cycle
  Other Names: Keytruda
Drug: Paclitaxel — Paclitaxel 80mg/m2 every 3 weeks by IV infusion on Days 1, 8, and 15 of each 3 week cycle
  Other Names: Taxol
  Arms: Arm A
Drug: Capecitabine — Capecitabine 2000mg every two weeks by mouth twice each day on days 1-7 of each 2 week cycle.
  Other Names: Xeloda
  Arms: Arm B

SUMMARY:
The goal of this study is to establish the safety and tolerability of pembrolizumab when administered in combination with either of two chemotherapy regimens (weekly paclitaxel or capecitabine) in unresectable/metastatic triple negative breast cancer (MTNBC) patients.

DETAILED DESCRIPTION:
In the pilot phase, patients will be enrolled to one of two experimental arms, which will be selected by the treating investigator (arm A: pembrolizumab + weekly paclitaxel; arm B: pembrolizumab + capecitabine).

Subjects will receive pembrolizumab via intravenous (IV) infusion at 200mg every three weeks (Q3W), and continue treatment Q3W until progression of disease, initiation of alternative cancer therapy, unacceptable toxicity, or other reasons to discontinue treatment occur, up to 24 months.

Paclitaxel will be administered intervenously on a weekly schedule at a dose of 80mg/m2.

Oral capecitabine will be administered at total daily dose of 4,000 mg (2,000 mg two times each day (abbreviated BID)). Capecitabine will be administered as intermittent therapy given on days 1-7 in 14-day cycles.

ELIGIBILITY:
Inclusion Criteria:

Be willing and able to provide written informed consent/assent for the trial.

* Be 18 years of age on day of signing informed consent.
* HER2-negative breast cancer (defined by immunohistochemistry (IHC) 0-1 (or) IHC 2 and in situ hybridization (ISH) HER2 / centromere on chromosome 17 (CEP17) < 2.0);
* ER and PR-negative breast cancer (defined by IHC<1%);
* Measurable metastatic or unresectable disease based on response evaluation criteria in solid tumours (RECIST) 1.1.
* Indicated for treatment with either weekly paclitaxel or oral capecitabine, as first or second-line chemotherapy in the metastatic/unresectable setting (as determined by the consenting investigator);
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained during screening. Archival tissue is acceptable if no intervening anti-neoplastic therapy has been administered, and if sufficient material is available for analysis (see section 8.0 for requirements);
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function as defined by protocol defined lab values
* Female subjects of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must avoid becoming pregnant while on treatment. Men must avoid fathering a child while on treatment.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study, Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. Denosumab is allowed.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with ≤ Grade 2 neuropathy and alopecia are an exception to this criterion and may qualify for the study.
* Has received the assigned chemotherapy regimen previously in the metastatic setting, or has received the assigned chemotherapy regimen previously in the (neo)adjuvant setting within 12 months of consent;
* If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that progressed or required active treatment in the last 5 years.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has history of/active pneumonitis requiring treatment with steroids or history of/active interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-programmed death 1 (anti-PD-1), anti-programmed death ligand 1 (anti-PD-L1), or anti-programmed death ligand 2 (anti-PD-L2) agent or has participated in a Merck-sponsored pembrolizumab study.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B or Hepatitis C.
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Page, MD, Principal Investigator — Medical Oncologist
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Providence Cancer Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Page DB, Pucilowska J, Chun B, Kim I, Sanchez K, Moxon N, Mellinger S, Wu Y, Koguchi Y, Conrad V, Redmond WL, Martel M, Sun Z, Campbell MB, Conlin A, Acheson A, Basho R, McAndrew P, El-Masry M, Park D, Bennetts L, Seitz RS, Nielsen TJ, McGregor K, Rajamanickam V, Bernard B, Urba WJ, McArthur HL. A phase Ib trial of pembrolizumab plus paclitaxel or flat-dose capecitabine in 1st/2nd line metastatic triple-negative breast cancer. NPJ Breast Cancer. 2023 Jun 21;9(1):53. doi: 10.1038/s41523-023-00541-2. PMID 37344474
- [Derived] Chun B, Pucilowska J, Chang S, Kim I, Nikitin B, Koguchi Y, Redmond WL, Bernard B, Rajamanickam V, Polaske N, Fields PA, Conrad V, Schmidt M, Urba WJ, Conlin AK, McArthur HL, Page DB. Changes in T-cell subsets and clonal repertoire during chemoimmunotherapy with pembrolizumab and paclitaxel or capecitabine for metastatic triple-negative breast cancer. J Immunother Cancer. 2022 Jan;10(1):e004033. doi: 10.1136/jitc-2021-004033. PMID 35086949
- See also: Providence Cancer Center — https://oregon.providence.org/our-services/p/providence-cancer-center/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Paclitaxel): pembrolizumab + weekly paclitaxel
  Pembrolizumab: Pembrolizumab 200mg every 3 weeks by IV infusion on Day 1 of each 3 week cycle
  Paclitaxel: Paclitaxel 80mg/m2 every 3 weeks by IV infusion on Days 1, 8, and 15 of each 3 week cycle
- Arm B (Capecitabine): pembrolizumab + capecitabine
  Pembrolizumab: Pembrolizumab 200mg every 3 weeks by IV infusion on Day 1 of each 3 week cycle
  Capecitabine: Capecitabine 2000mg every two weeks by mouth twice each day on days 1-7 of each 2 week cycle.
Period: Overall Study
Arm/Group | Arm A (Paclitaxel) | Arm B (Capecitabine)
Started | 15 | 14
Completed | 13 | 14
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Paclitaxel) | Arm B (Capecitabine) | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Customized [Mean (Standard Deviation); unit: years]
  Age, Mean (SD) | 56 (12.5) | 63 (8.7) | 59 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 9 | 13 | 22
  Non-Caucasian | 6 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29
ECOG Score [Count of Participants; unit: Participants] — Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; Grade 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; Grade 5: Dead
  Participants
    Grade 0 | 4 | 5 | 9
    Grade 1 | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Treatment-Associated Adverse Events Requiring Discontinuation
Description: The count of participants who experienced serious adverse events and grade III/IV treatment-associated adverse events requiring discontinuation of pembrolizumab.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Paclitaxel) | Arm B (Capecitabine)
Number analyzed (Participants) | 15 | 14
Participants
  Discontinued Patients | 2 | 0
  Continued Treatment | 13 | 14

2. Primary Outcome: Number of Patients Who Complete Chemotherapy Without a Dose Delay of More Than 21 Days.
Description: The number of patients who complete 6 weeks of chemotherapy without requiring a dose delay of more than 21 days.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Paclitaxel) | Arm B (Capecitabine)
Number analyzed (Participants) | 15 | 14
Participants
  Patients Completed Chemotherapy | 15 | 12
  Patients Requiring Dose Delay of More Than 21 Days | 0 | 2

3. Secondary Outcome: Overall Response Rate
Description: Patients will have a computerized tomography (CT) scan (preferred) or magnetic resonance imaging (MRI) scan at 12 weeks to measure the size of target lesions. The percentage of patients whose tumors respond to treatment at 12 weeks will be compared to historical controls. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR."
Time Frame: 12 weeks
Population: Two patients in Arm A discontinued from study at the 6 week mark and are not evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Paclitaxel) | Arm B (Capecitabine)
Number analyzed (Participants) | 13 | 14
percentage of participants | 31 [10 to 61] | 43 [18 to 71]

ADVERSE EVENTS:
Time Frame: ~21 weeks
Arm/Group | Arm A (Paclitaxel) | Arm B (Capecitabine)
All-Cause Mortality (participants affected / at risk) | 1/15 | 1/14
Serious Adverse Events (participants affected / at risk) | 5/15 | 4/14
Other Adverse Events (participants affected / at risk) | 15/15 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Paclitaxel) (N=15) | Arm B (Capecitabine) (N=14)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cancer Related Pain (General disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cardiac Arrest Resulting in Death (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Gram positive bacteremia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Liver failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Right hip fracture (femoral neck) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Syncope (Cardiac disorders) | 1 (1) | 0 (0)
Vasogenic edema (brain met) (General disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Worsening cancer pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Paclitaxel) (N=15) | Arm B (Capecitabine) (N=14)
Abdominal Cramping (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 3 (6)
Absolute neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Activated PTT prolonged (Investigations) | 0 (0) | 1 (1)
Acute encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Adhesive Capsulitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Amnesia (Psychiatric disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 7 (9) | 6 (15)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 7 (9)
Anxiety (Psychiatric disorders) | 2 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Edema, limbs (General disorders) | 5 (6) | 7 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bilateral tonsillar enlargement with erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Breast Pain (General disorders) | 0 (0) | 1 (1)
Breast tenderness (General disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 1 (1)
Common cold (General disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (5) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5)
Creatinine Increased (Investigations) | 0 (0) | 1 (2)
Cuticle pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (8) | 9 (21)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry desquamation (hand) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 4 (4)
Dry nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry scalp (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
DVT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 7 (8)
Ejection fraction decrease (Investigations) | 0 (0) | 1 (1)
Elevated AST (Investigations) | 0 (0) | 1 (1)
Elevated GGT (Investigations) | 0 (0) | 1 (1)
Elevated PTT (Investigations) | 0 (0) | 1 (1)
Emesis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema (General disorders) | 2 (2) | 1 (1)
Facial edema (General disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fatigue (General disorders) | 8 (9) | 9 (13)
Fever (General disorders) | 4 (5) | 4 (9)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 2 (3) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Fogginess (Psychiatric disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
GERD (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 2 (2)
Hand pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hand/Foot Syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 10 (21)
Headache (Nervous system disorders) | 0 (0) | 7 (9)
Hearing loss left ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (10)
Hypokalemia (Metabolism and nutrition disorders) | 5 (6) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (6) | 8 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 2 (6)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Increased Pain (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Jaw pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leg cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Loss of hand function (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Loss of voice (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (12)
Malaise (General disorders) | 0 (0) | 1 (1)
Melena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Memory loss (Nervous system disorders) | 0 (0) | 1 (1)
Mouth numbness (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mouth sores (Gastrointestinal disorders) | 1 (1) | 2 (3)
Mouth tenderness (Gastrointestinal disorders) | 2 (2) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail pain (General disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (12) | 8 (11)
Neck blisters (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Oral mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain, general (General disorders) | 5 (7) | 5 (7)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (9) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5)
Plugged Ears, Intermittent (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1)
Rash (any location) (Skin and subcutaneous tissue disorders) | 9 (12) | 2 (2)
Retching, Intermittent (Gastrointestinal disorders) | 1 (1) | 0 (0)
Right breast musculoskeletal episode (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rigors (General disorders) | 0 (0) | 1 (1)
Satiety (Gastrointestinal disorders) | 0 (0) | 1 (1)
Scratchy Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection, left breast (Infections and infestations) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Stye (eye infection) (Eye disorders) | 1 (1) | 0 (0)
Swollen neck lymph nodes (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Temple laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Transaminitis (Investigations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (2)
Urinary tract infection (Infections and infestations) | 2 (3) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal itch, Intermittent (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vision changes/disturbance (Eye disorders) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (4) | 4 (6)
Weight loss (Investigations) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
WBC decreased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT02734290/Prot_SAP_000.pdf